CLINICAL TRIAL: NCT00550485
Title: Blood-brain-barrier Permeability of Escitalopram Depending on Genetic Polymorphisms of the ABCB1-gene: Effect on Sleep and Procedural Learning
Brief Title: Pharmacokinetic and Pharmacodynamic Effects of Escitalopram Depending on Genetic Polymorphisms of the ABCB1-gene
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Max-Planck-Institute of Psychiatry (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: L3/2005
Record Dates: First submitted 2007-10-29; First posted 2007-10-30 (Estimated); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): Healthy subjects with a single nucleotide polymorphism (SNP) of the ABCB1-gene (Genotype A)
  Interventions: Drug: escitalopram
- 2 (Other): Healthy subjects with a single nucleotide polymorphism (SNP) of the ABCB1-gene (Genotype B)
  Interventions: Drug: escitalopram

INTERVENTIONS:
Drug: escitalopram — escitalopram 4 mg

SUMMARY:
The ABCB1-gene product P-glycoprotein is an integral membrane protein that actively transports substrates out of the intracellular compartment. One of the major sites of its action is the blood-brain-barrier. It is highly expressed in brain capillary endothelial cells and involved in limiting the access of substrates such as antidepressants to the central nervous system. A single nucleotide polymorphism (SNP) of the ABCB1-gene was recently identified showing a different treatment response to antidepressant drugs depending on the genotype. Therefore, it is assumed that healthy subjects with different genotypes of that SNP will be associated with significantly different brain levels of the antidepressant escitalopram after 6 days of intake. Sleep recordings are a useful bio-marker for effects of antidepressants on the CNS. Selective serotonin reuptake inhibitors (e.g. escitalopram) cause a suppression of REM sleep and a stronger fragmentation of sleep compared to untreated subjects. Higher plasma levels of antidepressants affected the sleep to a greater extent than lower levels. In line with this finding, we suppose that sleep EEG recordings of healthy subjects with different genotypes of the above mentioned SNP will be differently affected after taking 6 days escitalopram. In addition, effects of drug intake on the gene expression in lymphocytes and metabolic changes will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* healthy males 20-30 years

Exclusion Criteria:

* any medication

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2007-10; Primary Completion 2018-07-06 (Actual); Study Completion 2018-07-06 (Actual)

PRIMARY OUTCOMES:
Time spent in rapid-eye-movement (REM) sleep assessed by polysomnography. | after 6 days of intake of escitalopram
  Time spent in rapid-eye-movement (REM) sleep assessed by polysomnography.

SECONDARY OUTCOMES:
Sleep stages | after 6 days of intake of escitalopram
  Sleep stages beside REM sleep (wake, NonREM sleep) assessed by polysomnography
Sleep continuity | after 6 days of intake of escitalopram
  Sleep continuity measures assessed by polysomnography
ABCB1 gene expression | baseline and after 6 days of intake of escitalopram
  messenger ribonucleic acid (mRNA) expression of the target gene ABCB1
Metabolic changes | baseline and after 6 days of intake of escitalopram
  Small molecule metabolic changes in blood serum

CONTACTS AND LOCATIONS:
Overall Officials: Axel Steiger, MD, Principal Investigator — Max-Planck-Institute of Psychiatry
Locations (1):
- Max Planck Institute of Psychiatry, Munich, Germany